CLINICAL TRIAL: NCT02057471
Title: An Open Label Study of Intravenous Iron (FERINJECT) in Colorectal Adenocarcinoma Related Anaemia to Identify Potential Biomarkers of Responsiveness to Intravenous Iron
Brief Title: Intravenous Iron: Measuring Response in Anemic Surgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09GS002; 2009-011382-80 (EudraCT Number)
Record Dates: First submitted 2014-02-03; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Colorectal Neoplasm; Anemia
Keywords: Adenocarcinoma; Anemia; Blood Transfusion; Colorectal surgery; Preoperative care; Perioperative care; Postoperative care; Iron; Hematinics; Hepcidin; Quality of life; Postoperative complications
MeSH Terms: conditions — Colorectal Neoplasms; Anemia; Adenocarcinoma; Postoperative Complications | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Ferric Carboxymaltose (Experimental): All recruited patients will be allocated to this treatment. 1 gram of Ferric carboxymaltose (FERINJECT) to be given at recruitment
  Interventions: Drug: Intravenous ferric carboxymaltose

INTERVENTIONS:
Drug: Intravenous ferric carboxymaltose — 1 gram intravenous ferric carboxymaltose (FERINJECT) will be administered to all patients within the study
  Other Names: FERINJECT

SUMMARY:
20 Patients will be recruited with confirmed colorectal adenocarcinoma and anemia who are planned to undergo surgery. All patients will be treated with a single dose of 1g intravenous ferric carboxymaltose (FERINJECT).

It is hypothesized that intravenous iron supplementation is efficacious at raising haemoglobin levels and reduced blood transfusion requirements.

DETAILED DESCRIPTION:
Patients who are anemic at the time of operation have been shown to have an increased frequency of complications including wound infection and longer post-operative admissions. Similarly, patients who are anemic at the time of their cancer operation are more likely to require a blood transfusion which may increase the risk of recurrence of the cancer.

At present, oral iron is often used to treat anemia preoperatively in an attempt to minimize the risk above. This drug is often poorly tolerated due to the side effect profile. Blood transfusions can also be administered but expose the patient to other risks including infection and transfusion associated reactions. In order to overcome these issues, intravenous iron preparations have been developed and have improved in safety.

This is open label clinical trial, which looks to investigate the efficacy of intravenous iron is in the treatment of preoperative anemia in colorectal patients. The outcomes reviewed will include the amount and frequency of blood transfusions received, changes in patient blood profiles operative complications and hospital length of stay. The role of hepcidin as a biomarker of treatment response will also be assessed.

All data will be confidentially recorded on a Case Report Form, as will drug reactions and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosed with colonic or rectal adenocarcinoma
* Defined date of operation at least 14 days from recruitment to study
* Confirmed anemia
* Females of child bearing age must agree to use a medically accepted form of contraceptive

Exclusion Criteria:

* Patient's who are unable to consent
* Recognized allergy or intolerance of the study drug or excipients
* Patients with previous or current hematological disease that in the investigators' opinion would confound the diagnosis of anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of patients transfused allogenic red blood cells | Patients will be followed from recruitment to the study until postoperative discharge from hospital, which will be an expected average of 4 weeks
  To determine if the administration of intravenous iron reduces the number of expected allogenic red blood cell transfusions from recruitment to the perioperative phase
Hemoglobin levels | Patients will be followed from recruitment to the study until 8 weeks post operatively, which will be an expected average of 10 weeks
  To determine if intravenous iron significantly increases hemoglobin levels in the preoperative optimization of patients

SECONDARY OUTCOMES:
Hepcidin levels | Patients will be followed from recruitment to the study until the day after surgery, which will be an expected average of 3 weeks
  To monitor changes in hepcidin in response to treatment and review if this can predict response to intravenous iron therapy
Erythropoietin levels | Patients will be followed from recruitment to the study until 8 weeks post operatively, which will be an expected average of 10 weeks
  To monitor changes in Erythropoietin in response to treatment and review if this can predict response to intravenous iron therapy
Transferrin saturation levels | Patients will be followed from recruitment to the study until 8 weeks post operatively, which will be an expected average of 10 weeks
  To monitor changes in transferrin saturation levels in response to treatment and review if this can predict response to intravenous iron therapy
Ferritin levels | Patients will be followed from recruitment to the study until 8 weeks post operatively, which will be an expected average of 10 weeks
  To monitor changes in ferritin levels in response to treatment and review if this can predict response to intravenous iron therapy
C Reactive Protein levels | Patients will be followed from recruitment to the study until 8 weeks post operatively, which will be an expected average of 10 weeks
  To monitor changes in C Reactive Protein levels over the course of the study, and review if this can predict response to intravenous iron therapy, or is associated with changes in hepcidin

OTHER OUTCOMES:
Number of adverse events associated with intravenous iron infusion | Patients will be followed from recruitment to the study until postoperative discharge from hospital, which will be an expected average of 4 weeks
  To assess the safety and feasibility of the principle of administration of intravenous iron in a single dose, preoperative outpatient visit

CONTACTS AND LOCATIONS:
Overall Officials: Austin G Acheson, MD FRCS, Study Chair — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom